CLINICAL TRIAL: NCT07213817
Title: An Open-Label, Phase I/II First-in-Human, Dose Escalation, Dose Optimisation and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetic, Pharmacodynamic, Immunogenicity and Antitumour Activity of IPN60300 as Single Agent in Adult Participants With Locally Advanced or Metastatic Solid Tumours.
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetic, Pharmacodynamic, Immunogenicity and Antitumour Activity of IPN60300 in Adults With Locally Advanced or Metastatic Solid Tumours
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-60300-450
Record Dates: First submitted 2025-10-01; First posted 2025-10-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Part 1a is sequential assignment - non-randomized, single arm. Part 1b is randomized, two-arm, parallel design.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase Ia: Dose escalation (Experimental): IPN60300 will be administered at assigned dose level.
  Interventions: Biological: IPN60300
- Phase Ib : Dose optimisation (Experimental): Participants will be randomised to one of the two doses of interest.
  Interventions: Biological: IPN60300

INTERVENTIONS:
Biological: IPN60300 — IPN60300 will be administered at assigned dose level.

SUMMARY:
This study aims to find the right dosage and evaluate the safety and effectiveness of the drug IPN60300 in adults with advanced solid tumours, which are cancers that have spread to other parts of the body from their original location. All participants will receive the drug by injection.

Study Phases:

* Phase Ia: Participants with certain types of tumours will be treated in cohorts of increasingly higher doses of the drug to determine the safe and effective dose range (a high and a low dose).
* Phase Ib: Participants with a specific tumour type will receive one of the two doses identified in phase Ia. The dose level will be assigned randomly (by chance).

Study Periods:

Screening: Up to 28 days before first IPN60300 injection to determine eligibility.

Treatment: Starts with the first dose of IPN60300 and continues until it needs to be stopped due to harmful effects, the disease getting worse, or if the participant decides to stop taking part in the study, the investigator's decision to stop treatment, death or the study is terminated early by the sponsor.

Participants will undergo blood tests, urine collections, physical examinations, and clinical evaluations.

ELIGIBILITY:
Inclusion criteria:

* Participant must be ≥18 years of age, at the time of signing the informed consent.
* Participants with histologically or cytologically documented, locally advanced, or metastatic solid tumors, that relapsed or were refractory after being previously treated with standard of care therapy; or for which there is no available established therapy; or standard therapy is contraindicated or not deemed appropriate by the treating investigator.
* Participants must have measurable disease per Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Male and female participants Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Adequate bone marrow function within 7 days before first dose of study intervention,
* Adequate renal function within 7 days before first dose of study intervention,
* Adequate hepatic function or laboratory abnormalities indicating hepatic injury within 7 days before first dose of study intervention,
* Prothrombin time or international normalised ratio (INR) ≤1.5 × ULN.
* At the time of screening, a tumour tissue specimen is required for enrolment into the dose escalation and dose optimisation portions of the study for retrospective central laboratory determination.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).
* Have a life expectancy of more than 3 months for disease-related mortality, as evaluated by the investigator.

Exclusion Criteria:

* Known second malignancy either progressing or requiring active treatment within the last 2 years prior to first dose of study intervention.
* Residual toxicity from prior anticancer therapy that are NCI CTCAE version 5.0 Grade 2 or higher. Stable chronic Grade 2 toxicities from previous treatments may be eligible per the judgement of investigator.
* History of major surgery within 4 weeks prior to the first dose of study intervention.
* Previous solid organ transplantation.
* Pre-existing, acute or chronic severe corneal disorders, sequelae from severe corneal disorders, or a history of corneal transplantation.
* Active brain metastases or leptomeningeal metastases with exception to asymptomatic and treated brain metastases (i.e. no neurological symptoms, no requirements for corticosteroids and lesions <1.5 cm), which are stable and not expected to become symptomatic in the next 3 months in the opinion of the investigator.
* History of stroke or significant cerebrovascular disease (ie, transient ischemic attack) within 6 months prior to initiation of study intervention.
* History of clinically significant cardiac disease within 6 months prior to the initiation of study intervention, including but not limited to unstable angina, acute myocardial infarction, endoscopic or open-heart cardiac surgery, or heart failure classified as New York Heart Association Grade 2 or higher.
* History of clinically significant respiratory disease within 6 months prior to the initiation of study intervention, including severe chronic obstructive pulmonary disease or asthma.
* History of noninfectious interstitial lung disease (ILD)/pneumonitis/radiation pneumonitis that required steroids or has current ILD/pneumonitis.
* Clinically significant gastrointestinal disorder including bleeding, occlusion, diarrhoea >Grade 1, malabsorption syndrome, ulcerative colitis, inflammatory bowel disease or partial bowel obstruction.
* Any evidence of severe active infection or inflammatory condition.
* Significant concurrent, uncontrolled medical condition that would put participants at unacceptable risk from study participation or preclude them from complying with study procedures as per investigator assessment, including, but not limited to renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral, or psychiatric disease.
* Participants with uncontrolled human immunodeficiency virus (HIV). HIV infected participants are eligible if they meet criteria described in the protocol.
* Known active infection with hepatitis B virus (HBV) OR hepatitis C virus (HCV). Participants are eligible if they meet criteria described in the protocol.
* Ongoing immunosuppressive therapy, including systemic corticosteroids. NOTE: Physiologic replacement or use of topical or inhaled corticosteroids are allowed.
* Concurrent participation in another therapeutic treatment trial, previous participation should respect the minimum of 5 half-lives or 4 weeks before the study intervention initiation (whichever is shorter).
* Participants accommodated in an institution because of regulatory or legal order; prisoners or participants who are legally institutionalised.
* For French participants only: participants are under court protection, not affiliated to a social security system or protected adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Percentage of participants with dose limiting toxicity (DLT) | within 21 days following study drug administration.
Phase Ia and Ib: Percentage of participants experiencing Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TE SAEs). | From the first IPN60300 administration until 30 days after the last dose
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A TEAE is an AE for which the start date is on or after the date that the intervention began or it was present prior to receiving the intervention but the intensity increased during the active phase of the study.
Phase Ib: Objective response rate (ORR) | At end of study (up to approximately 3 years )
  ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR), as determined by investigator per RECIST version 1.1

SECONDARY OUTCOMES:
Phase Ia: Time to maximum observed drug concentration (tmax) of IPN60300 after single and multiple doses of IPN60300 | within 21 days following study drug administration
Phase Ia: Maximum observed drug concentration (cmax) of IPN60300 after single and multiple doses of IPN60300 | Within 21 days following study drug administration
Phase Ia: Area under the plasma concentration time curve over one dosing interval (AUCtau) of IPN60300 after single and multiple doses of IPN60300 | Within 21 days following study drug administration
Phase Ia: Tmax of Total Antibody after single and multiple doses of IPN60300 | Within 21 days following study drug administration.
Phase Ia: Cmax of Total Antibody after single and multiple doses of IPN60300 | Within 21 days following study drug administration.
Phase Ia: AUCtau of Total Antibody after single and multiple doses of IPN60300 | Within 21 days following study drug administration.
Phase Ia: Tmax of free toxin after single and multiple doses of IPN60300 | Within 21 days following study drug administration.
Phase Ia: Cmax of free toxin after single and multiple doses of IPN60300 | Within 21 days following study drug administration.
Phase Ia: AUCtau of free toxin after single and multiple doses of IPN60300 | Within 21 days following study drug administration.
Phase Ia and Ib: Percentage of Treatment-Emergent Anti-Drug Antibodies (ADA), Including Binding and Neutralizing Antibodies. | Prior study drug administration until the End of Treatment (EoT) visit (approximately up to 3 years
Phase Ia: Objective Response Rate (ORR) | At end of study (up to approximately 3 years)
  ORR is defined as the percentage of participants with BOR of CR or PR, as determined by investigator per RECIST version 1.1
Phase Ib: Duration of response (DoR) | At end of study (up to approximately 3 years)
  DoR is defined as the time from the first documented evidence of CR or PR until progressive disease, as determined by investigator per RECIST version 1.1, or death from any cause, whichever occurs first
Phase Ib: Progression-free survival (PFS) | At end of study (up to approximately 3 years)
  PFS is defined as the time from the date of first IPN60300 administration to the date of the first documented disease progression, as determined by investigator per RECIST version 1.1, or death due to any cause, whichever occurs first
Phase Ib: Disease control rate (DCR) | At end of study (up to approximately 3 years)
  DCR is defined as the percentage of participants with BOR of CR, PR or stable disease (SD), as determined by investigator per RECIST version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (12):
- United States (6):
  - Yale Cancer Center-Yale University, New Haven, Connecticut
  - START Midwest, Grand Rapids, Michigan
  - Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - NEXT Oncology, Fairfax, Virginia
- France (3):
  - Centre Leon Berard, Lyon
  - Institut de Cancerologie de l'Ouest (ICO)- CRLCC Rene Gauducheau, Saint-Herblain
  - Gustave Roussy Cancer Campus Grand Paris- (Institut de Cancerologie Gustave-Roussy), Villejuif
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - NEXT Quiron-Barcelona, Barcelona
  - START Madrid CIOCC Hospital Universitario HM Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/